CLINICAL TRIAL: NCT02456415
Title: A Prospective, Single Center, Single Group, Open-label Study to Evaluate the Efficacy and Safety of Magnesium Alloy Screw as a Novel Bioabsorbable Material in Patients Requiring Internal Fixation Due to Hand Fractures
Brief Title: The Efficacy and Safety of Magnesium Alloy Screw as a Novel Bioabsorbable Material in Patients Due to Hand Fractures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U&I Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNI-01
Record Dates: First submitted 2015-05-15; First posted 2015-05-28 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-05

CONDITIONS: Hand Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- K-MET™ Bioresorbable Bone screw (Experimental): The K-MET™ Bioresorbable Bone Screw, intended to be used for trauma therapy, consists of Cortex screws, Cannulated headless screws. For Headless screw and Cannulated headless screws, the design is similar to normal headless compression screws but the compression function was achieved by using different lengths for the front and rear pitches. These screws are dynamic and allow therewith the fracture at the Carpal, metacarpal, and small hand bone.
  Interventions: Device: K-MET™ Bioresorbable Bone screw

INTERVENTIONS:
Device: K-MET™ Bioresorbable Bone screw — The biodegradable screw inserted into bone with an appropriate driver is slowly degraded and is completely degraded after completion of bone union and absorbed into the body. The screw is indicated for fixing damaged bone.

SUMMARY:
This study evaluates the safety and efficacy of biodegradable magnesium alloy screw, in patients with hand fractures who require internal fixation (to obtain a product license from the Ministry of Food and Drug Safety in Korea (MFDS)).

DETAILED DESCRIPTION:
Rationale: Hand fractures including intra- and extra-articular phalanges and metacarpal are common and account for approximately 40% of upper extremity fractures and lead to functional loss of the hand.Fractures can be treated conservatively with a nonsurgical approach(Closed reduction) by placing the damaged figure in a splint; this may results in displacement, rotation, angulation and/or instability, therefore require surgery. Surgical techniques for treatment of hand fractures include internal fixation with metal plate or screws after Open reduction and external fixation with insertion of percutaneous pins or screws. Percutaneous external fixation is one of the widely used methods, but is difficult to maintained when accompanied by unstable fractures and soft tissue injuries or there are severely comminuted fractures and sometimes results in restricted motion of adjacent joints due to prolonged fixation. In comparison, internal fixation is an operation using internal fixators such as plates, wires, screws etc. solely or concurrently depending on the location and severity of hand fracture. With the recent advancement of implant design and fixation techniques, a variety of screws are widely used for fixation of small-bone fractures.

The present study was designed to evaluate the efficacy and safety of magnesium alloy screw as a novel bioabsorbable and biodegradable material.

Study Duration: After an approval of clinical protocol from MFDS in Korea, total 20 months were required including 14 months for subject enrollment and 6 months of follow-up. An additional 1 month was required after completion of the study for handling of data, statistical analysis and preparation of study report.

Target Subjects: Patients who require internal fixation using screws due to hand fractures

Investigational Device: K-MET™ Bioresorbable Bone screw (manufactured by U&I) This device divided into two type,Cortex screw and Headless compression screw.

Number of Subjects: A total of 34 cases of bone fractures in 28 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 20 years or older
* Patients who require internal fixation using screws in the hand
* The clinical features of hand fractures are oblique and spiral fractures
* Patients who voluntarily submitted a written informed consent and are willing to and able to follow the clinical study protocol.

Exclusion Criteria:

* Infections around the fracture site or soft-tissue injury greater than Grade III
* Fracture patterns such as open, transverse or comminuted fracture with greater than type II
* Fractures that require the use of wires, pins or plates for fixation
* Patients with re-fracture
* Patients with critical systemic diseases
* Patients with renal failure showing plasma creatinine level exceed 1.4 at the screening
* Pregnant, lactating women
* Patients who have a history of allergy to magnesium alloy
* Patients with presence of past illness or taking a drug that may affect bone union
* Patients who have participated in other clinical study and treated with medication or other medical device within past 3 months
* Patients who are judged not to be appropriate for study enrollment in the opinion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Bone union | up to 6 months
  Bone union was evaluated at 6-month after surgery according to the following definition.Definition of bone union is when simple X-ray findings reveal that bone trabeculae or cortical bone exceeds the fracture site. Non-union is defined as no union at 3-month post-surgery.

SECONDARY OUTCOMES:
PROM(Passive Range of Motion) | up to 6 months
  This Passive Range of Motion(PROM) is measured by goniometer and is compared with the value of the normal hand that did not undergo surgery.
TAM(Total Active Motion) | up to 6 months
  Total Active Motion(TAM) is measured by goniometer and is compared with the value of the normal hand that did not undergo surgery.
Power(grip strength and pick-up power) | up to 6 months
  The Power was measured using a dynamometer and pick-up counter and is compared with the value of the hand that did not undergo surgery.
DASH scale | 3,6 months
  This questionnaire evaluates the ability of the hand to perform certain activities before and after surgery. It was directly completed by subjects.
Pain as measured by the NRS (1~10) | up to 6 months
  The NRS (1~10) was used to measure the level of pain and was compared before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gyeong-jin Han, professor, Principal Investigator — Ajou Univ hospital